CLINICAL TRIAL: NCT06200948
Title: Effects of Aerobic Cycling Training in Patients With Gynecologic Cancer-related Lower Extremity Lymphedema: A Randomized Comparative Study
Brief Title: Effects of Aerobic Cycling Training in Patients With Gynecologic Cancer-related Lower Extremity Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Onur Kara, Medical Doctor (Physical Medicine and Rehabilitation Resident Doctor), Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10025140
Record Dates: First submitted 2023-12-08; First posted 2024-01-11 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Lymphedema; Lymphedema, Lower Limb; Gynecologic Cancer
Keywords: Aerobic training; Cycling ergometry; Gynecological cancer; Lymphedema
MeSH Terms: conditions — Lymphedema | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: While the patients in non-cycling group will get only complete decongestive treatment (CDT) for 3 weeks, the patients in cycling group will get CDT+cycling ergometry treatment for 3 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-cycling group (Active Comparator): patients will receive only complete decongestive treatment
  Interventions: Other: Complete Decongestive Treatment
- cycling group (Active Comparator): patients will receive complete decongestive treatment + cycling ergometry treatment
  Interventions: Other: Aerobic Exercise; Other: Complete Decongestive Treatment

INTERVENTIONS:
Other: Aerobic Exercise — While the patients in non-cycling group will get only complete decongestive treatment (CDT) for 3 weeks, the patients in cycling group will get CDT+cycling ergometry treatment for 3 weeks. Cycling ergometry treatment will be performed with Voit AT-200 Black Collection horizontal bike for 20 minutes. Exercise intensity will be adjusted to %40-59 of heart rate reserve (HRR).
  Arms: cycling group
Other: Complete Decongestive Treatment — While the patients in non-cycling group will get only complete decongestive treatment (CDT) for 3 weeks, the patients in cycling group will get CDT+cycling ergometry treatment for 3 weeks. Cycling ergometry treatment will be performed with Voit AT-200 Black Collection horizontal bike for 20 minutes. Exercise intensity will be adjusted to %40-59 of heart rate reserve (HRR).

SUMMARY:
Comparison of complete decongestive treatment and complete decongestive treatment + cycling ergometry treatment in patients with gynecologic cancer-related lower extremity lymphedema in terms of quality of life, lower extremity functionality and lower extremity volume measurement

DETAILED DESCRIPTION:
After being informed about study and potential risks, all patients giving written informed consent will undergo screening period determine eligibility for study entry. The patients who met the eligibility recruitments will get into the assessment.

The study will include 63 participants (31 controls and 32 interventions). Simple randomization will be preferred in this study. The coin toss method will be used for simple randomization.

Researcher will record demographic and clinical data of the patients and will evaluate the patients' pre-treatment volumes by circumference measurement method. Researcher will evaluate quality of life by lymphedema quality of life questionnaire (LYMQOL) and lower extremity functionality by lower extremity functional scale (LEFS). While the patients in non-cycling group will get only complete decongestive treatment (CDT) for 3 weeks, the patients in cycling group will get CDT+cycling ergometry treatment for 3 weeks.Cycling ergometry treatment will be performed with Voit AT-200 Black Collection horizontal bike for 20 minutes. Exercise intensity will be adjusted to %40-59 of heart rate reserve (HRR). At the end of treatment; Researcher will evaluate volume, functionality and quality of life of the patients again and will compare the two groups in terms of volume measurement, functionality and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Being cognitively competent
* Chemotherapy radiotherapy etc. treatment has been completed and there is no oncological risk
* Signing written informed consent to participate in the study

Exclusion Criteria:

* Cardiac failure
* Uncontrolled hypertension
* Having kidney failure
* Having a systemic infection
* Local infection such as erysipelas and cellulitis in the lower extremities
* Venous insufficiency (DVT etc.)
* Presence of any neuromuscular disease affecting the lower extremities
* Having lipolymphedema
* Fracture in the lower extremity
* Having active metastasis
* Having a language problem
* Being pregnant
* Being unable to continue treatment

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Effect of Aerobic Training | baseline and at 3rd weeks
  Assesment of the effect of aerobic training on quality of life, functionality and volume difference in patients with gynecologic cancer-related lower extremity lymphedema

CONTACTS AND LOCATIONS:
Overall Officials: Onur Kara, M.D., Principal Investigator — Health Sciences University, Ankara Bilkent City Hospital; Gül Mete Civelek, M.D., Study Director — Health Sciences University, Ankara Bilkent City Hospital; Meltem Dalyan, M.D., Study Chair — Health Sciences University, Ankara Bilkent City Hospital; Cansu Şahbaz Pirinççi, Pt. (PhD.), Study Chair — Health Sciences University, Gulhane Physiotherapy and Rehabilitation Faculty; Rabia Tarlabölen, Pt., Study Chair — Health Sciences University, Ankara Bilkent City Hospital
Locations (1):
- Ankara Bilkent City Hospital Physical Therapy and Rehabilitation Hospital, Ankara, Bilkent/Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kendrova L, Mikulakova W, Urbanova K, Andrascikova S, Zultakova S, Takac P, Peresta Y. Comprehensive Decongestive Therapy as a Treatment for Secondary Lymphedema of the Lower Extremity and Quality of Life of Women After Gynecological Cancer Surgery. Med Sci Monit. 2020 Jun 17;26:e924071. doi: 10.12659/MSM.924071. PMID 32555125
- [Result] Dionne A, Goulet S, Leone M, Comtois AS. Aquatic Exercise Training Outcomes on Functional Capacity, Quality of Life, and Lower Limb Lymphedema: Pilot Study. J Altern Complement Med. 2018 Sep/Oct;24(9-10):1007-1009. doi: 10.1089/acm.2018.0041. PMID 30247973
- [Derived] Kara O, Mete Civelek G, Sahbaz Pirincci C, Tarlabolen R, Dalyan M. Effects of aerobic cycling training in patients with gynaecologic cancer-related lower extremity lymphedema: A randomised comparative study. Support Care Cancer. 2025 Mar 19;33(4):302. doi: 10.1007/s00520-025-09354-4. PMID 40108020
- See also: Comprehensive Decongestive Therapy as a Treatment for Secondary Lymphedema of the Lower Extremity and Quality of Life of Women After Gynecological Cancer Surgery — https://pubmed.ncbi.nlm.nih.gov/32555125/
- See also: Aquatic Exercise Training Outcomes on Functional Capacity, Quality of Life, and Lower Limb Lymphedema: Pilot Study — https://pubmed.ncbi.nlm.nih.gov/30247973/